CLINICAL TRIAL: NCT04640246
Title: A Phase 1/2 Multi-Center Dose-Escalation Study of the Safety, Tolerability and Early Efficacy of TBX-3400 in Subjects With Solid Malignant Tumors Resistant or Refractory to Standard Therapies
Brief Title: Study of TBX-3400 in Subjects With Solid Malignant Tumors Resistant or Refractory to Standard Therapies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taiga Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBX-3400-003
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Cancer; Tumor, Solid; Refractory Cancer
Keywords: Cancer; Solid tumor; Malignant; Refractory; Resistant
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TBX-3400 (Experimental): TBX-3400 by intravenous infusion
  Interventions: Biological: TBX-3400

INTERVENTIONS:
Biological: TBX-3400 — Autologous transfusion

SUMMARY:
This is a study of treatment with TBX-3400 in subjects with solid malignant tumors that are resistant or refractory to standard therapies.

The subject's own blood cells are exposed to a protein that has been shown in the laboratory to result in anti-tumor activity.

The study hypothesis is that TBX-3400 cells will enhance anti-tumor activity and improve the body's immune response to the tumor.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in the study:

1. Histologically or cytologically confirmed diagnosis of malignant solid tumor/s
2. Male or female subjects age 18 or older
3. Metastatic tumor that has failed at least one line of therapy with further options being non-curative; or with metastatic tumor and patient declines standard of care therapies and alternatives offered, at the discretion of the investigator
4. At least 28 days or 5 half-lives, since the last dose of medication to treat their malignancy.
5. Measurable or evaluable disease by RECIST version 1.1
6. Capable of understanding and complying with protocol requirements
7. A life expectancy of greater than 12 weeks at Screening
8. ECOG Performance Status of 0 to 2
9. Written informed consent from the patient or the patient's legally acceptable representative prior to the initiation of any study procedures
10. Adequate bone marrow, liver, and renal function at screening as defined below:

    * hemoglobin ≥8.0 g/dL (transfusions allowed)
    * total lymphocyte count ≥500/µL
    * absolute neutrophil count ≥1500/µL
    * platelet count ≥100,000/µL (transfusions allowed)
    * alanine transaminase and aspartate transaminase ≤3.0 times the upper limit of normal (ULN), or ≤5 times ULN for subjects with known hepatic metastases
    * total serum bilirubin ≤1.5 x the ULN; ≤2.0 x the ULN if liver metastases are present; subjects with a known history of Gilbert's syndrome (≤3.0 x the ULN) and/or isolated elevations of indirect bilirubin are eligible for study participation
    * estimated glomerular filtration rate ≥50 mL/min/1.73 m2 (using Cockcroft Gault formula)

Exclusion Criteria:

Subjects who meet any of the following criteria will not be eligible for participation in the study:

1. Pregnant or breast feeding
2. Require systemic pharmacologic doses of corticosteroids at or above the equivalent of 10 mg/day of prednisone; replacement doses, topical, ophthalmologic and inhalational steroids are permitted
3. Active, symptomatic central nervous system (CNS) metastases. Subjects with CNS metastases are eligible for the trial if the metastases have been treated by surgery and/or radiotherapy and the patient is off corticosteroids and is neurologically stable for at least 7 days prior to screening and the Medical Monitor approves subject inclusion
4. Any concurrent uncontrolled illness, including mental illness or substance abuse, which in the opinion of the investigator would make the patient unable to cooperate or participate in the trial
5. Severe uncontrolled cardiac disease within 3 months of study entry, including unstable or new onset angina, myocardial infarction or cerebrovascular accident
6. Women of child-bearing potential who are unable or unwilling to use an acceptable method of contraception
7. Known infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C (in USA: Known infection with human immunodeficiency virus [HIV], hepatitis B or hepatitis C that is not controlled and has any related symptoms)
8. Symptomatic congestive heart failure, defined as New York Heart Association Class II or higher
9. Systemic lupus erythematous (SLE), inflammatory bowel disease, primary Sjogren's syndrome, rheumatoid arthritis, systemic sclerosis, and granulomatosis with polyangiitis; and any other autoimmune condition that, in the opinion of the investigator, may increase the risk of trial participation or trial drug administration, unless reviewed and approved by the medical monitor.
10. Any hematopoietic malignancy
11. Have more than one primary cancer diagnosis within the last 3 years
12. Organ transplant or requiring immune suppression
13. Bullous pemphigoid and other autoimmune diseases of the dermal-epidermal junction; these include bullous pemphigoid, bullous SLE, liner IgA disease, epidermolysis bullosa acquisita, and other pemphigoid variants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the incidence and severity of treatment-emergent adverse events (TEAEs), including the incidence of dose-limiting toxicities (DLTs), graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. | 8 months
  Adverse events from subject reporting

SECONDARY OUTCOMES:
Tumor Responses as defined by RECIST | 8 months
  Tumor measurements to assess disease state
Assessment of concentrations of certain proteins such as cluster of differentiation 69 (CD69), as biomarkers of activity of TBX-3400 | 8 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Presence and/or concentration of anti TBX-3400 antibodies | 8 months
  Measure of immunogenicity of TBX-3400

OTHER OUTCOMES:
Quantification of the concentration of interleukin-1 (IL-1) in plasma | 8 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Quantification of the concentration of interleukin-6 (IL-6) in plasma | 8 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Quantification of the concentration of interferon-alpha (IFN-α) in plasma | 8 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Quantification of the concentration of interferon-gamma inducible protein 10kD (IP-10) in plasma | 8 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Quantification of the concentration of interferon-gamma (IFN-γ) in plasma | 8 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Quantification of the concentration of transforming growth factor-beta (TGF-ß) in plasma | 8 months
  Preliminary efficacy assessment to measure activity of TBX-3400

CONTACTS AND LOCATIONS:
Locations (2):
- The Angeles Clinic and Research Institute, Los Angeles, California, United States
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No